CLINICAL TRIAL: NCT02298504
Title: Evaluation of MTA Pulpotomy, Biodentine Pulpotomy, and Glass Ionomer Indirect Pulp Treatment in Primary Teeth
Brief Title: Vital Pulp Treatment in Primary Teeth
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Vineet Dhar, Associate Professor, Graduate Program Director, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-00058711
Record Dates: First submitted 2014-11-14; First posted 2014-11-24 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Vital Pulp Therapies; Indirect Pulp Cap; Pulpotomy
MeSH Terms: interventions — mineral trioxide aggregate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Indirect pulp cap (Experimental): IDP will be performed for this group
  Interventions: Device: Vitrebond
- MTA pulpotomy (Experimental): MTA pulpotomy will be performed for this group
  Interventions: Drug: Mineral Trioxide Aggregate
- Biodentin pulpotomy (Experimental): Biodentin pulpotomy will be performed for this group
  Interventions: Drug: Biodentin

INTERVENTIONS:
Drug: Mineral Trioxide Aggregate — Vital pulp therapy
  Other Names: MTA pulpotomy
  Arms: MTA pulpotomy
Drug: Biodentin — Vital pulp therapy
  Other Names: Biodentin Pulpotomy
  Arms: Biodentin pulpotomy
Device: Vitrebond — Vital pulp therapy
  Other Names: Indirect pulp cap
  Arms: Indirect pulp cap

SUMMARY:
In primary teeth, decay that is near the pulp (tooth nerve)is treated with either a pulpotomy or indirect pulp treatment if the tooth is not going to be extracted A pulpotomy involves removing the top 1/2 of the pulp, placing a medication/material on the pulp, covering the remaining pulp with a cement, and the restoring the tooth. The purpose of this pilot study is to gain preliminary information regarding the success of Biodentine, MTA, and IPT in the treatment of deep decay in children's primary molars.

DETAILED DESCRIPTION:
Pediatric patients having deep decay in primary molars seen at UMMC, UMSOD, and University of Maryland Rehabilitation and Orthopaedic Institute, will be included in the sample. Teeth with deep caries, >50% into dentin, will be randomly assigned using a table of random numbers to the three treatment groups:

Group 1 pulpotomy with MTA, Group 2 pulpotomy with Biodentine, Group 3 indirect pulp treatment. Treatment will be performed by board certified pediatric dentists or they will directly supervise pediatric dental residents at each site as part of their regular protocol for treating deep caries.

Radiographs will be taken as prescribed in the Guideline for taking Radiographs in Children by the American Academy of Pediatric Dentistry.

Twice yearly clinical examinations will be performed by the treating dentists or pediatric dental residents to check for any soft tissue pathology such as abscess or mobility of treated tooth/teeth. If treatment success/failure consensus between the blinded dentists is not reached, a third dentist will be consulted.

The success/failure data will be entered onto spreadsheets and examined statistically using statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with deep dental decay in primary molars
* Teeth with signs and symptoms of reversible pulpitis

Exclusion Criteria:

* Teeth with clinical symptoms of irriversible pulpitis or pulp necrosis or acute dental infection
* Children with systemic illness that contraindicated vital pulp treatment such a sickle cell disease
* Teeth that are not restorable

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success after pulpotomy | 3 years
  No signs of abscess or any swelling related to the tooth, no signs of fistula or other pathology, no signs of pathologic mobility, no post-operative pain, no pain on palpation or percussion of the tooth
Clinical success after indirect pulp cap | 3 years
  No signs of abscess or any swelling related to the tooth, no signs of fistula or other pathology, no signs of pathologic mobility, no post-operative pain, no pain on palpation or percussion of the tooth
Radiographic success after pulpotomy | 3 years
  No signs of root resorption (internal or external), no signs of furcation involvement or periapical radiolucency, no signs of loss of lamina dura, presence of normal appearance of periodontal ligament space

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Dentistry, Baltimore, Maryland, United States